CLINICAL TRIAL: NCT00659919
Title: Treatment of Neuroleptic Induced Acute Akathisia With Trazodone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BeerYaakov Mental Health Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Trazodone-60CTIL
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): The patients in this arm received placebo
  Interventions: Drug: Placebo
- Trazodone (Active Comparator): The patients on this arm received Trazodone for 3 consecutive days
  Interventions: Drug: Trazodone

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Trazodone
  Arms: Trazodone

SUMMARY:
Administration of trazodone for the treatment of neuroleptic induced acute akathisia in a cross-over fashion of 6 days duration. 3 days of placebo and 3 days of trazodone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with akathisia according to DSM-IV criteria at least mild akathisia.

Exclusion Criteria:

* Change of pharmacologic regimen 7 days prior to study entry
* Significant systemic disease
* The presence of chronic akathisia
* Patients unable to cooperate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2000-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Barnes Akathisia rating scale, Positive and Negative syndrome scale, Hamilton Depression Rating Scale, Hamilton Anxiety Scale, Clinical Global Impression, Scale for the Assessment of Negative Symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Beer Yaakov MHC, Beer Yaacov, Israel